CLINICAL TRIAL: NCT04474119
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Phase III Study to Assess the Efficacy and Safety of KN046 Combined With Platinum-containing Chemotherapy Versus Placebo Combined With Platinum-containing Chemotherapy in First Line Advanced Squamous Non-small Cell Lung Cancer Subjects (ENREACH-L-01)
Brief Title: KN046 in Subjects With Advanced Squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KN046-301
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Squamous Non-small-cell Lung Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): KN046 plus Carboplatin and Paclitaxel
  Interventions: Drug: KN046
- Control arm (Placebo Comparator): Placebo plus Carboplatin and Paclitaxel
  Interventions: Drug: KN046 placebo

INTERVENTIONS:
Drug: KN046 — In combine therapy stage, KN046 is 5 milligram per kilogram, every 3 weeks. In maintain stage, KN046 is 5 milligram per kilogram, every 2 weeks.
  Arms: Experimental arm
Drug: KN046 placebo — In combine therapy stage, KN046 placebo is 5 milligram per kilogram, every 3 weeks.
  In maintain stage, KN046 placebo is 5 milligram per kilogram, every 2 weeks.
  Arms: Control arm

SUMMARY:
This study is a randomized, double-blind, multicenter, phase III clinical study to compare the clinical efficacy and safety of KN046 plus paclitaxel and carboplatin versus placebo plus paclitaxel and carboplatin in subjects with advanced squamous NSCLC who have not previously received systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-confirmed or cytologically confirmed diagnosis of stage IV squamous NSCLC.
* No known epidermal growth factor receptor (EGFR) mutations.
* Has measurable disease.
* Has not received prior systemic treatment for their advanced/metastatic NSCLC.
* Can provide tumor tissue.
* Has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function
* If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment;
* If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment.

Exclusion Criteria:

* Untreated active CNS metastasis or leptomeningeal metastasis.
* Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first dose of trial treatment;
* Has received other anti-tumor treatment within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first trial treatment;
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment;
* Curative radiation within 3 months of the first dose of trial treatment. Radiation to more than 30% of the bone marrow or with a wide field of radiation should not be used within 4 weeks prior to the first administration of trial treatment;
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids);
* Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines);
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;
* History or current active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Previous malignant disease
* History of uncontrolled intercurrent illness
* Prior therapy with any antibody/drug targeting T cell coregulatory proteins
* Known severe hypersensitivity reactions to antibody drug
* Is pregnant or breastfeeding;
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Blinded Central Imaging | up to 2 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.
Overall Survival (OS) | up to 3 years
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Investigators | up to 2 years
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No